CLINICAL TRIAL: NCT06069921
Title: Ultrasound-based Deep Learning Signature and Radiomics Signature Nomogram for Diagnosis of Benign and Malignant Breast Lesions of BI-RADS Category 4 Using Intratumoral and Peritumoral Regions
Brief Title: Using Deep Learning and Radiomics to Diagnose Benign and Malignant Breast Lesions Based on Ultrasound
Status: Completed | Type: Observational
Sponsor: Ma Zhe (Other)
Responsible Party: Sponsor-Investigator, Ma Zhe, Director of Ultrasound, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Other Study IDs: YXLL-KY-2023(045)
Record Dates: First submitted 2023-09-29; First posted 2023-10-06 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Breast Diseases
MeSH Terms: conditions — Breast Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- maligant: female patients with US-visible solid maligant breast masses who underwent biopsy and/or surgical resection.
- benign: female patients with US-visible solid benign breast masses who underwent biopsy and/or surgical resection.

SUMMARY:
This retrospective study aimed to create a prediction model using deep learning and radiomics features extracted from intratumoral and peritumoral regions of breast lesions in ultrasound images, to diagnose benign and malignant breast lesions with BI-RADS 4 classification.

Materials and methods: Patients who visited in The First Affiliated Hospital of Shandong First Medical University ＆ Shandong Provincial Qianfoshan Hospital were collected. Their general clinical features, information on preoperative ultrasound diagnosis, and postoperative pathologic data were reviewed.

ELIGIBILITY:
Inclusion Criteria:

* female patients with US-visible solid breast masses who underwent biopsy and/or surgical resection, and were classified as having BI-RADS 4 lesions in medical US reports.

Exclusion Criteria:

* preoperative endocrine therapy, chemotherapy, or radiotherapy, preoperative invasive breast operation, insufficient image quality, and no pathological results.

Ages: 15 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with breast lesions attending the First Affiliated Hospital of Shandong First Medical University were selected.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
radiomcis prediction model and the model evaluation | Immediately evaluated after the radiomcis prediction model was built
  three radiomics models were established using the support vector machines algorithm based on features extracted from the intratumoral, peritumoral, and combined regions of the breast lesions.The models were evaluated using various metrics, including AUC, accuracy, sensitivity, specificity, PPV, and NPV

SECONDARY OUTCOMES:
deep learning prediction model and the model evaluation | Immediately evaluated after the deep learning prediction model was built
  three deep learning models were established using the support vector machines algorithm based on features extracted from the intratumoral, peritumoral, and combined regions of the breast lesions.The models were evaluated using various metrics, including AUC, accuracy, sensitivity, specificity, PPV, and NPV

OTHER OUTCOMES:
the combination prediction model and the model evaluation | Immediately evaluated after the combination prediction model was built
  the combination model was established using clinical features , deep learning score and radiomics score.The models were evaluated using various metrics, including AUC, accuracy, sensitivity, specificity, PPV, and NPV

CONTACTS AND LOCATIONS:
Locations (1):
- QianfoshanH, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No
Lack of resources or infrastructure: Sharing IPDs requires resources and infrastructure to ensure data security, manage access requests and provide necessary documentation. Currently these resources are not well developed, so it may be difficult to share IPDs.